CLINICAL TRIAL: NCT02413320
Title: Randomized Open Label Phase II Trial of Neoadjuvant Carboplatin Plus Docetaxel or Carboplatin Plus Paclitaxel Followed by Doxorubicin Plus Cyclophosphamide in Stage I-III Triple-negative Breast Cancer
Brief Title: Neoadjuvant Study of Two Platinum Regimens in Triple Negative Breast Cancer
Acronym: NeoSTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Priyanka Sharma (Other)
Responsible Party: Sponsor-Investigator, Priyanka Sharma, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-IIT-Neoadjuvant-BRST-TNBC
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Triple-negative Breast Cancer
Keywords: TNBC, breast cancer, neoadjuvant, carboplatin, docetaxel, paclitaxel, doxorubicin, cyclophosphamide
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin + Paclitaxel then Doxorubicin + Cyclophosphamide (Active Comparator): Paclitaxel (80mg/m2) given IV every week x12 weeks and Carboplatin (AUC 6) given IV every 21 days x 4 cycles, followed by Doxorubicin (60mg/m2) given IV and Cyclophosphamide (600mg/m2) given IV every 14 days X 4 cycles
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin; Drug: Cyclophosphamide
- Carboplatin + Docetaxel (Active Comparator): Carboplatin (AUC 6) given IV and Docetaxel (75mg/m2) given IV every 21 days x 6 cycles
  Interventions: Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: taxol
  Arms: Carboplatin + Paclitaxel then Doxorubicin + Cyclophosphamide
Drug: Carboplatin
  Other Names: paraplatin
Drug: Doxorubicin
  Other Names: adriamycin
  Arms: Carboplatin + Paclitaxel then Doxorubicin + Cyclophosphamide
Drug: Cyclophosphamide
  Other Names: cytoxin, procytox
  Arms: Carboplatin + Paclitaxel then Doxorubicin + Cyclophosphamide
Drug: Docetaxel
  Other Names: taxotere
  Arms: Carboplatin + Docetaxel

SUMMARY:
Evaluate if the two carboplatin containing chemotherapy regimens will reduce the growth of breast cancer cells in women with Stage I, II, or III triple negative breast cancer.

DETAILED DESCRIPTION:
Sporadic and germline BRCA mutation associated triple-negative breast cancer share several pathological and molecular similarities which have led to the exploration of DNA damaging agents like platinum compounds in patients with triple-negative breast cancer. Recent studies demonstrate that addition of neoadjuvant carboplatin to doxorubicin/cyclophosphamide/taxane-based chemotherapy improves pathological complete response in patients with stage I-III triple-negative breast cancer but also increase toxicity.

A recent study reported encouraging pathological complete response rates with a non-anthracycline carboplatin plus docetaxel neoadjuvant chemotherapy regimen in a cohort of 49 triple negative breast cancer patients. This chemotherapy regimen of carboplatin plus docetaxel yielded an overall pathological complete response rate of 65% in unselected triple-negative breast cancer with pathological complete response rates of 61% in sporadic and 77% in germline BRCA-associated triple-negative breast cancer. The chemotherapy regimen of carboplatin/docetaxel is well tolerated and should be studied further and compared with regimens that add carboplatin to the standard anthracycline/taxane containing regimens.

This is the basis for the proposed randomized neoadjuvant phase II study to further estimate and compare pathological complete response rates of carboplatin plus docetaxel x 6 cycles to carboplatin plus paclitaxel x 4 cycles followed by doxorubicin plus cyclophosphamide x 4 cycles in stage I-III triple negative-breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage I (T>1cm), II or III triple negative breast cancer who have not had definitive breast surgery or received systemic chemotherapy
* The invasive tumor must be hormone receptor-poor, defined as both estrogen receptor and progesterone receptor staining present in ≤ 10% of invasive cancer cells by Immunohistochemistry.
* HER- 2 negativity will be based on the current ASCO-CAP guidelines for HER testing
* No prior chemotherapy, endocrine therapy or radiation therapy with therapeutic intent for this cancer
* Female subjects age 18 - 70 years
* ECOG Performance Status of 0-1
* Adequate organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/uL
  * Absolute neutrophil count ≥ 1500/uL
  * Platelets ≥ 100,000/uL
  * Total bilirubin ≤ 1.5mg/dL
  * AST(SGOT)/ALT(SPGT) ≤ 2 x institutional upper limit of normal
  * Creatinine ≤ 1.5mg/dl and/or Creatinine Clearance ≥ 60mL/min
  * Serum albumin ≥ 3.0 g/dL
* Women of child-bearing potential must agree to use adequate contraception
* Pretreatment lab values must be performed within 14 days of treatment initiation, and other baseline studies performed within 30 days prior to registration
* Subjects should have LVEF ≥ 50% by echocardiogram or MUGA scan performed within 4 weeks prior to treatment initiation
* Subjects should have breast and axillary imaging with breast MRI or breast and axillary ultrasound within 4 weeks prior to treatment initiation
* Subjects with clinically/radiologically abnormal axillary lymph nodes should have pathological confirmation of disease with image guided biopsy/fine needle aspiration.
* Subjects must be already enrolled in P.R.O.G.E.C.T observational registry
* Staging to rule out metastatic disease is recommended for subjects with clinical stage III disease
* Subjects with bilateral disease are eligible if they meet other eligibility criteria.
* Neuropathy: No baseline neuropathy grade > 2

Exclusion Criteria:

* Current or anticipated use of other investigational agents
* Subject has received chemotherapy, radiotherapy or surgery for the treatment of breast cancer
* Subject with metastatic disease
* History of allergic reactions to compounds of similar chemical or biologic composition to carboplatin, docetaxel, doxorubicin, cyclophosphamide, paclitaxel, or other agents used in the study
* Subjects with inflammatory breast cancer
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Subject is pregnant or nursing
* Subjects with concomitant or previous malignancies within the last 5 years. Exceptions include: adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and ductal carcinoma in situ (DCIS).
* Ejection Fraction <50% on ECHO or MUGA
* Cardiac function: Subjects with congestive heart failure, myocardial infarction, unstable angina pectoris, an arterial thrombotic event, stroke or transient ischemia attack within the past 12 months, uncontrolled hypertension (Systolic BP>160 or Diastolic BP>90), uncontrolled or symptomatic arrhythmia, or grade ≥ 2 peripheral vascular disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-07; Primary Completion 2019-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — University of Kansas Medical Center
Locations (9):
- United States (9):
  - University of Kansas Cancer Center - CRC, Fairway, Kansas
  - Hays Medical Center, Hays, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri

REFERENCES:
- [Result] Sharma P, Kimler BF, O'Dea A, Nye L, Wang YY, Yoder R, Staley JM, Prochaska L, Wagner J, Amin AL, Larson K, Balanoff C, Elia M, Crane G, Madhusudhana S, Hoffmann M, Sheehan M, Rodriguez R, Finke K, Shah R, Satelli D, Shrestha A, Beck L, McKittrick R, Pluenneke R, Raja V, Beeki V, Corum L, Heldstab J, LaFaver S, Prager M, Phadnis M, Mudaranthakam DP, Jensen RA, Godwin AK, Salgado R, Mehta K, Khan Q. Randomized Phase II Trial of Anthracycline-free and Anthracycline-containing Neoadjuvant Carboplatin Chemotherapy Regimens in Stage I-III Triple-negative Breast Cancer (NeoSTOP). Clin Cancer Res. 2021 Feb 15;27(4):975-982. doi: 10.1158/1078-0432.CCR-20-3646. Epub 2020 Nov 18. PMID 33208340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide | Carboplatin + Docetaxel
Started | 49 | 52
Completed | 48 | 52
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide | Carboplatin + Docetaxel | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Median (Full Range); unit: years] | 51 [32 to 69] | 54 [29 to 70] | 51 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 36 | 71
  Black or African American | 9 | 10 | 19
  Asian | 2 | 1 | 3
  Other | 2 | 5 | 7
  Hispanic | 1 | 1 | 2
  Non-Hispanic | 47 | 51 | 98
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 100
Lymph node status [Count of Participants; unit: Participants]
  Negative | 34 | 36 | 70
  Positive | 14 | 16 | 30
T stage [Count of Participants; unit: Participants] — Primary tumor stage, as defined by the 7th edition of the American Joint Committee on Cancer's staging manual. T stage indicates the size or extent of the primary tumor. T1: tumor ≤20 mm in greatest dimension; T2: tumor >20 mm but ≤50 mm in greatest dimension; T3: tumor >50 mm in greatest dimension; T4: tumor of any size with direct extension to the chest wall and/or to the skin (ulceration or skin nodules).
  Participants
    T1 | 11 | 8 | 19
    T2 | 31 | 39 | 70
    T3-4 | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathological Complete Response
Description: To evaluate the pathological complete response rates with neoadjuvant chemotherapy regimens of carboplatin plus paclitaxel x 4 cycles followed by doxorubicin plus cyclophosphamide X 4 cycles and carboplatin plus docetaxel X 6 cycles in subjects with stage I-III triple-negative breast cancer. Pathological complete response is defined as no evidence of disease in the breast and axilla at the time of pathology review except for DCIS.
Time Frame: 20 weeks
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide | Carboplatin + Docetaxel
Number analyzed (Participants) | 48 | 52
Participants | 26 | 28

2. Secondary Outcome: Number of Participants With Minimal Residual Disease
Description: To evaluate minimal residual disease rates (residual cancer burden 0+1) with two neoadjuvant chemotherapy regimens in subjects with stage I-III triple-negative breast cancer.
Time Frame: 20 weeks
Population: Patients with residual cancer burden index available
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide | Carboplatin + Docetaxel
Number analyzed (Participants) | 46 | 52
Participants | 31 | 35

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Adverse events (serious and non-serious) of grade 3 or 4, definitely related/probably related/possibly related to study treatment, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Patients were systematically evaluated for toxicity at each visit.
Arm/Group | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide | Carboplatin + Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 41/48 | 13/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin + Paclitaxel Then Doxorubicin + Cyclophosphamide (N=48) | Carboplatin + Docetaxel (N=52)
Anemia (Blood and lymphatic system disorders) | 22 | 2
Neutropenia (Blood and lymphatic system disorders) | 29 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 0
Hypokalemia (Investigations) | 2 | 1
Hyponatremia (Investigations) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 4
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Infection (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT02413320/Prot_SAP_000.pdf